CLINICAL TRIAL: NCT05493449
Title: Impact of School Milk Program on Nutritional, Body Composition and School Performance of Primary School Children in Attock and Sheikhupura
Brief Title: Impact of School Milk Program on Nutritional Status of Primary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Collaborators: University of Lahore (Other); Friesland campina Engro Pakistan (Unknown)
Responsible Party: Principal Investigator, Sanaullah Iqbal, Associate Professor, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: School Milk Program
Record Dates: First submitted 2022-06-20; First posted 2022-08-09 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Milk Intervention on Body Composition and School Attendance

STUDY DESIGN:
Intervention Model Description: There were three groups in study. Group A is the one which received UHT Milk, Group B received Flavored Milk and Group C was a control group.
Masking Description: No masking is involved as participants, investigator and assessor know intervention types
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): In this group, no milk (intervention) was provided
- UHT Milk (Experimental): In this group, UHT Milk intervention was provided
  Interventions: Combination Product: UHT Milk
- Flavored Milk (Experimental): In this group, flavored milk was provided to participants
  Interventions: Combination Product: Flavored Milk

INTERVENTIONS:
Combination Product: UHT Milk — In this group of participants, UHT milk, 180 mL was provided and results were compared with control and flavored milk group
  Arms: UHT Milk
Combination Product: Flavored Milk — In this group of participants, flavored milk, 180 mL was provided and results were compared with control and UHT group
  Arms: Flavored Milk

SUMMARY:
Malnutrition is very common in Pakistan, especially in children of under developed areas due to lack of resources and access to nutritious food. It can disturb the normal physical and mental development as well as functioning in children which can put economic burden on country level.

Therefore, school meal programs can play an important role in providing school children with healthy and nutritious food which can improve their nutritional status as well as overall health.

DETAILED DESCRIPTION:
The proposed intervention study was conducted in the primary school going children of age 4-16 years old in two districts of Punjab namely Attock and Sheikhpura with collaboration of University of Veterinary and Animal Sciences, Lahore, University of Education, Lahore and Friesland Campina (Engro Foods Pvt. Ltd.), Pakistan. The participants of study was students studying in classes nursery to 5, out of study population of 90 Schools of different tehsils of two districts (Attock city and Sheikupura city), Punjab-Pakistan that are being run by the administration of University of Education, Lahore.

The study participants for research are 8.9 % of 7799 total population involved in school milk program children i.e. total 693 (380 Attock city and 313 Sheikhupura). A total of 18 schools (9 from each district) was selected as a sample of the study population, since there were three groups (A-Group to receive Full Cream Milk; B-Group to receive Flavored Milk; C-Group is control) and three schools in each districts form each group. In addition, the selected schools have been selected in each district in a way in both selected districts to have a uniform population of around 160±5.

At initiation of the study, baseline data was collected from the study participants. Data regarding socio-demographic factors, 24-hrs dietary recall, anthropometric, school attendance, body composition, dietary deficiency signs and symptoms was collected from study population i.e. 693 students. After baseline findings, for dietary intervention, the sample population based on schools was divided into 3 clusters/group including control, Ultra High Temperature (UHT) and flavored milk as intervention groups (i.e., UHT and flavored milk groups, were given milk (180 mL/participants/day; on alternate days basis and/or daily basis as the case may be owing to Covid situation) for 3 months. The data was collected from study participants at different intervals initiation (baseline) and termination (3 months), whereas, data after 2 months of termination will be collected to estimate washout period differences of the intervention on the study parameters. After the completion of study, the control group will also receive milk for same duration on humanitarian basis.

Inclusion Criteria: Children having no symptoms of Lactose Intolerance Exclusion Criteria: Children having symptoms of Lactose Intolerance

Informed Consent and other considerations:

All the protocols of study were explained to study participants/teachers and informed consent was obtained prior to enrollment in the study. The data was considered as relevant and reliable, if 70% of the sample (compared to start of the study) completes the study with minimum of 80% of allocated milk consumption. If any student(s) wants to quit during the course of the study, he/she do it on his/her will and was not forced to complete the study.

Data Analysis:

Descriptive analysis was carried out by using SPSS version 25 (SPSS for windows version 25; SPSS Inc., Chicago, IL, USA), Microsoft excel and World Health Organization Anthroplus (Software) was used to calculate height for age and BMI for age z scores. The data was analyzed by using independent sample t-test, paired sample t-test and one-way ANOVA, statistical significance was at p > 0.05.

ELIGIBILITY:
Inclusion Criteria:

• Participants aged 4-16 years of age enrolled under University of Education, Lahore who are having no symptoms of Lactose Intolerance

Exclusion Criteria:

• Participants having symptoms of Lactose Intolerance

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7799 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Weight | change from baseline to 3 months
  Weight of the study participants was measured by using weighing balance.
Height | change from baseline to 3 months
  Height of the study participants was measured by using stadiometer.
Total Body Water (TBW) | change from baseline to 3 months
  TBW of the study participants was measured by using body composition analyzer Inbody J-270.
Body Protein | change from baseline to 3 months
  Body protein of the study participants was measured by using body composition analyzer Inbody J-270.
Minerals | change from baseline to 3 months
  Body minerals of the study participants was measured by using body composition analyzer Inbody J-270.
Body Fat Mass (BFM) | change from baseline to 3 months
  Body fat mass of the study participants was measured by using body composition analyzer Inbody J-270.
Skeletal Muscle Mass (SMM) | change from baseline to 3 months
  SMM of the study participants was measured by using body composition analyzer Inbody J-270.
Percentage Body Fat (PBF) | change from baseline to 3 months
  PBF of the study participants was measured by using body composition analyzer Inbody J-270.
Inbody Score | change from baseline to 3 months
  Inbody Score of the study participants was measured by using body composition analyzer Inbody J-270.
Visceral Fat Level (VFL) | change from baseline to 3 months
  VFL of the study participants was measured by using body composition analyzer Inbody J-270.
Waist to Hip ratio (WHR) | change from baseline to 3 months
  WHR of the study participants was measured by using body composition analyzer Inbody J-270.

SECONDARY OUTCOMES:
Attendance percentage | change from baseline to 3 months
  Student attendance from school records was evaluated for documenting their involvement and performance.
Nutritional deficiency Assessment | change from baseline to 3 months
  The study participants were examined physically to check nutritional deficiencies along with signs & symptoms including hair, mouth, lips, eyes, gums, teeth, tongue, face, skin, nails, musculoskeletal and neck etc.
  Deficiencies related to various macro and micronutrients were also examined i.e., energy, proteins, vitamin A, D, calcium, riboflavin, Vitamin B12 etc.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Veterinary and Animal Sciences, Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No